CLINICAL TRIAL: NCT03522766
Title: Evaluation of Urine Samples and Their Relation to Urinary Tract Infection
Status: Completed | Type: Observational
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CP287
Record Dates: First submitted 2018-05-01; First posted 2018-05-11 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy volunteers with no urinary tract infections: people who don't experience urinary tract infections
  Interventions: Other: urine sample
- Healthy volunteers with urinary tract infections: people who frequently experience urinary tract infections
  Interventions: Other: urine sample
- Intermittent catheter users with neurogenic bladder
  Interventions: Other: urine sample
- Intermittent catheter users with enlarged prostate
  Interventions: Other: urine sample

INTERVENTIONS:
Other: urine sample — The subjects are asked to give a maximum of 15 urine samples during the study

SUMMARY:
The aim is to explore the human urine composition and its relation to urine tract infections

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. For the 2 patient populations: Use intermittent catheter on a daily basis due to neurogenic bladder or enlarged prostate and have used IC for at least 2 months
4. For healthy volunteers without UTIs: No diag-nosed UTIs within the last year
5. For healthy volunteers with recurrent UTIs: 3 or more UTIs within the last year or 2 UTIs within the last 6 months (treated with antibiotics)

Exclusion Criteria:

1. Be treated for urinary tract infection at time of enrolment
2. May not take prophylactic treatment for urinary tract infections (antibiotics only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of danish subjects and will consist of healthy volunteers as well as users of intermittent catheter (neurogenic bladder or enlarged prostate) with and without reoccurring urine tract infections.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Type of bacteria present in the urine | 1 year
  The different bacteria isolated present in the urine will be identified

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, PhD, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark